CLINICAL TRIAL: NCT02527356
Title: Advancing Mobility and Socialization in Toddlers With Disabilities: a Trial to Assess the Effects of Modified Toy Cars Training With Different Postures
Brief Title: Advancing Mobility and Socialization in Toddlers With Disabilities: Modified Toy Cars Training With Different Postures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MOST-104-2314-B-182-023-MY3
Record Dates: First submitted 2015-08-17; First posted 2015-08-19 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2019-07

CONDITIONS: Children With Mobility Disabilities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ROC-Stand group (Experimental): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for ride-on car with standing posture training (ROC-stand).
  Interventions: Behavioral: Ride-On Cars with Standing Posture (ROC-Stand)
- ROC-Sit group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for ride-on car with standing posture training (ROC-sit)
  Interventions: Behavioral: Ride-On Cars with Standing Postures (ROC-Sit)
- Regular Therapy group (Active Comparator): The participant's performance is indicative of the extent to which early power mobility training is feasible for 1 to 3 years old and diagnosed as motor delay (>1.5 sd). Parents/caregivers and occupational therapists will be responsible for regular therapy.
  Interventions: Behavioral: Regular Therapy Program

INTERVENTIONS:
Behavioral: Ride-On Cars with Standing Posture (ROC-Stand) — The 2-hour training session is composed of two 30-minute driving sessions and two 25-minute natural play sessions, with a 10-minute break. Every week's treatment program will be before planned and adjusted by the therapist and the caregivers through discussion and clinical observation of participant's performance in the previous session. Training will concentrate on building the concept of casual-effect on the switch and car motion, goal-oriented driving in a hospital, and upper limb use in functional tasks with driving and hand use in functional tasks for exploration in natural play session.
  Arms: ROC-Stand group
Behavioral: Ride-On Cars with Standing Postures (ROC-Sit) — Most of the guidelines are similar with ROC-Stand, except for the posture of driving. The training time and period is the same as ROC-Stand. The two 30-minute driving sessions can also be divided into 4 times of 15-minute sessions, depending on the child's standing ability with supported condition.
  Arms: ROC-Sit group
Behavioral: Regular Therapy Program — The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS). The regular therapy group will continue the regular therapy, including physical, occupational and speech therapy. In addition, they will receive training program in a hospital for 2 hours/per session, 2 sessions/per week for a total of 12-week intervention. The participants will also experience the two 30-minute car driving sessions during the whole 2-hour training. The difference between the regular therapy group and the two ROC groups is the experience of car driving is controlled by the therapist, i.e. passive locomotion. The general propose of the training is to improve the developmental scales, mobility, socialization and upper limb use in functional tasks. The research team will videotape the child's natural play and driving performance for 1 hour/per session, 1 session/per week during the 12-week intervention phase.
  Arms: Regular Therapy group

SUMMARY:
The three purposes of this study are: 1) to examine the feasibility and effects of ride-on car training with two different postures on mobility and socialization in toddlers with disabilities; 2) to quantify whether toddlers with disabilities are able to have more exploratory behaviors and social interactions with ride-on car training through observation and wrist-worn accelerators; 3) to determine the critical factors of using the different modes of modified ride-on toy car on family perceptions and participation.

The concept of using modified ride-on toy cars (ROC) in therapy has became a novel application in recent years. This study is further to examine the effects of ride-on toy car training with two different postures, i.e., sitting and standing , on independent mobility, exploration and socialization through low-cost, family-centered approach. It will also improve family's understanding of children's capabilities, which improves their development. Based on the power analysis from the preliminary results of investigator group study, investigators will recruit 60 children with disabilities who are between 1 to 3 years old and diagnosed as motor delay. They will be randomly assigned to one of the following three groups: ROC-Sit group, ROC-Stand group and regular therapy group. The whole study duration will be 24 weeks, including 12-week intervention and 12-week follow-up; the total amount of treatment will be equal for three groups. Standardized assessments are provided for a total of three times during the study, including the time before and after the intervention and in the end of the follow-up phase. The ROC-Sit and ROC-Stand programs will be administered by the therapist and include 120 minutes/per session, 2 sessions/per week. The research team will visit the hospital once/per week to provide 60 minutes videotaping and let participants wear wrist-worn accelerators. The regular therapy group will continue their regular therapy without any additional car driving training. The research team will visit them once/per week for the assessments. The assessments include standardized measurements and behavioral coding from the videotapes and accelerators. The findings of this study will provide a novel therapeutic tool (i.e., combining the low-tech modified ride-on cars with different postures) on advancing children's mobility, socialization, family participation and development.

DETAILED DESCRIPTION:
Pediatric rehabilitation, through training and assistive technology (AT), seeks to provide children with disabilities with the same level of mobility, exploration, socialization and participation for children with typical development (TD). There are many basic barriers to achieving this high standard and no single AT or combination of AT can currently provide the level of mobility and exploration that children, families and therapists desire. Currently, the most critical barrier to including power mobility in EI programs is the lack of readily available power chairs for children younger than 2-3 years of age, the period when mobility is rapidly developing for children with TD. Certain characteristics of the most common commercial pediatric power wheelchairs limit their use in the home and community spaces such as playgrounds. These limitations include price, size and weight, transportation requirements, maintenance, aesthetics and social acceptance. Experimental power mobility devices (PMD) have the potential to address some of these limitations such as size, weight and infant use. Unfortunately these are likely years from commercial availability. Moreover, power wheelchairs have historically been designed to address a limited set of goals related to mobility with minimal consideration of socialization. Although of increasing interest, there is very little empirical evidence of the effects or even feasibility of early power mobility training on overall development and the family participation, particularly for socialization. Investigator believe there is a need for readily available mobility options for immediate use by very young children and their families that address some of the above limitations while expanding the role of PMD past simply mobility and into socialization.

In this study, investigator will modify two types of modified ride-on cars (ROCs) for toddlers with disabilities for the use in clinical settings as part of a 24-week power mobility training program. In addition, investigator will compare the effects of applying early power mobility training to the regular therapy on development. Investigator will focus on four research questions. Specifically, can investigator: 1) use the modified toy cars with two different postures as effective power mobility training programs to improve the independent mobility and socialization; 2) select a set of dependent measures that quantify whether the children increase their exploratory and social behaviors; 3)conduct a hospital-based, power mobility training program that results in a high level of fun for the child and compliance by the family and therapists. In addition, investigator will examine whether the effects of increased independent mobility and socialization will affect toddler's function with the 3 International Classification of Function (ICF) domains. If investigator results are generally positive and show significant differences on independent mobility and socialization among the early power mobility training programs with two different postures and regular therapy, it will provide us some alternative ways to advance independent mobility and socialization. Subsequently, the further randomized controlled trial studies can quantify the effectiveness and the feasibility with different treatment intensity and various pediatric populations.

The specific aims of this study are: 1) to examine the feasibility and effects of ROC training with two different postures on mobility and socialization in toddlers with disabilities; 2) to quantify whether toddlers with disabilities are able to have more exploratory behaviors and social interactions with ROC training through observation and wrist-worn accelerometers; 3) to determine the critical factors of using the different modes of modified ROC on family perceptions and participation. Through the comparison among the two ROC training groups (i.e., treatment groups) and regular therapy group (i.e., control group), investigator hypothesize that both groups of ROC training will have more improvements on functional mobility, socialization and parenting stress than the control group. Specifically, the treatment group of ROC training with standing posture will have more increased social function than the sitting posture in the ROC training and control group. In addition, toddlers in both treatment groups will have more physical activity for exploration, in comparison with the control group. Investigator also hypothesize that ROC training with different postures will elicit different family perceptions on the child's capabilities and themselves, i.e., caregivers, in comparison with the regular therapy.

Study Design: A multiple group pretest-posttest control group design will be applied. Three groups will be involved in this project: ride-on car with sitting posture (ROC-Sit), ride-on car with standing posture (ROC-Stand) and regular therapy. The participants will be randomly assigned to one of the three groups by using the well-sealed, opaque envelopes when they are recruited in the study. Once the participants are recruited in the study, the research team will modify a toy car based on each participant's group and capabilities during this pre-intervention phase (the first two or three weeks before intervention starts), e.g., seat and steering wheel modifications. All the modifications can be disassembled so they can be adjusted based on each participant's progress during the intervention. The study duration for each participant is 24-week, including 12-week intervention and 12-week follow-up.

Participants in the study will be 60 infants or preschool children ages 12 months to 36 months with motor delays (sd > 1.5). The age group of infants/preschool children was selected based on the previous studies on early power mobility training in infants and preschool children.

Recruitment: The children will be recruited from self-referrals, health care practitioners, or the hospitals in Taipei and Taoyuan, Taiwan where children with motor delays (>1.5 sd) are receiving outpatient rehabilitation. The research team will initially post flyers describing the study at clinical settings and contacted the therapists in the clinical settings to introduce the goals,criteria and general procedure of the study. Parents/guardians will obtain information about the study through the flyers and their therapists. When the research team contacts the parents, study will be explained and parents will receive a letter detailing the procedure and given an opportunity to ask questions. Parents/guardians will sign this informed consent form at the time of the first visit.

Procedure: Before the pre-intervention assessments, the research team will modify the car's seat and acceleration to the hand switch-driven, which allows the car to be derivable for the participant who meets the inclusion criteria. Each participant of the ROC training groups will have either a customized, sitting-style toy car or a standing-style toy car, depending on the assigned group. In addition to the original design of the sitting-style toy car in investigator previous studies, investigator have added the seat height, extra seat belts and pipe frame to ensure the participant's safety and the whole device's stability during the standing mode of locomotion. After modifications, they will receive pre-intervention assessments, including behavioral videotaping and developmental assessments. The developmental assessments will occur at the first and last week of the 12-week intervention, and the end of the 12-week follow-up phase. A therapist who does not involve in the intervention and is blinded to the study purpose will complete all the developmental tests. The driving and socialization behaviors will be videotaped by the research team for 1 hour/per session, 1 session/per week before, during and after the intervention phase at the hospital. In addition, participants will wear two accelerometers on their wrists to monitor the physical activity during the 1 hour videotaping session. All videotapes will be coded by two independent coders, who are undergraduate students. Prior to making their ratings, the coder is instructed as to coding procedures by the PI, but he/she is not informed about the group assignment and the purpose of the study.

Intervention The research team will ask caregivers to identify goals (before intervention), and measure progress using goal-attainment scaling (GAS) before and after the intervention for the three groups. All three groups will continue their regular therapy during the intervention phase. Each group will receive the ROC training or the conventional therapy for 2 sessions/per week during this phase. The ROC training includes driving the ROC with a sitting or a standing posture based on the ecological and dynamic systems theories. The regular therapy group will receive additional conventional therapy based on the developmental and motor learning theories.

Follow-up This period will focus on the 12-week follow-up after receiving a treatment program. No treatment programs will be delivered to the participants. The research team will still videotape the child's natural play and driving performance at the hospital for 1 hour /per session, 1 session/per week during the 12-week follow-up phase.

Data Reduction and Analysis All videotapes will be coded by two independent coders, who are undergraduate students. Prior to making their ratings, the coder is instructed as to coding procedures, but he/she is not informed about the group assignment and the purpose of the study.

From the 1 hour filmed session during intervention, each participant's 20 'most active' minutes of 2 training play sessions (i.e., 10 minutes of driving and 10 minutes of natural play) are selected for coding. Thus, the 20-minute 'most-active' minutes are categorized as 10-minute 'Car Play' (from driving training) and 10-minute 'Natural Play'. Mobility Measures The behavioral measures were obtained via video coding the 10-minute Car Play during pre-intervention, intervention and post-intervention phases to determine the feasibility of learning to drive the car.

Repeated measure one way ANOVA will be used to compare the mean difference of using different toy cars on mobility, socialization and exploratory behaviors before and after the intervention, and after 12-week follow-up, i.e., within group comparison. One way ANOVA will be used to compare the mean difference of all developmental tests, participation and physical activity for exploration among three groups before and after the intervention and the end of follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Motor delays resulting in motor impairments that prevented independent walking (standard deviation (SD) < -1.5, assessed by the Chinese Child Development Inventory (CCDI) via a pediatric physician) )
2. Able to stand independently for 2 seconds or to tolerate standing with support for 10 minutes
3. Able to reach the objects with either one or two hands
4. The height is between 69 to 103 cm and the weight is between 7-18 kg
5. Consent of the parents to agree to the testing procedures and participate in the training program

Exclusion Criteria:

1. Children with severe sensory impairments such as blindness, deafness
2. The height is not between 69 to 103 cm and the weight is not between 7 to 18 kg
3. Parents/caregivers are not able to make a time commitment for the training phase.

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2015-11-05 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in General Mobility and Social Development at 12 weeks and 24 weeks as assessed by the Pediatric Evaluation of Disability Inventory (PEDI) | Assessment will occur 3 times during the whole study, including the first and last week of the 12-week intervention, and the end of the 12-week follow-up phase
  PEDI is a set of tests for children from 8 months to 6 years old. The PEDI quantified self-care, mobility, and social functions. The PEDI is especially useful for tracking changes in functional skills.
Mobility/Driving Performance as assessed by the coding behaviors from the videotaping | The driving behaviors will be followed for the duration of implementing the intervention and follow-up program at the hospital, an expected average of 24 weeks.
  The driving behaviors were coded from each 10-minute Car Play session: a) amount of time moving/total time, b) frequency, time and duration of parental assistance (physical and/or vocal), c) number of successful "directional driving trials". In each of 10 trials, the child is asked to drive 5 feet to the parent or researcher. He/she is given 30 seconds to complete the distance and make a stop at the goal.
Socialization as assessed by the coding behaviors from the videotaping | The socialization behaviors will be followed for the duration of implementing the intervention and follow-up program at the hospital, an expected average of 24 weeks.
  The frequency and duration related to socialization will be coded during the whole 20-minute Play, including 10-minute Natural Play and 10-minute Car Play: physical contacts, initiation of contact with others, other initiated contacts, facial expressions, vocalizations/gestures and mutual play events (ex. sharing a toy).
Physical Activity for Exploration as assessed by the number of counts recorded from the accelerators wearing on both wrists | The physical activity for exploration behavior will be followed for the duration of implementing the intervention and follow-up program at the hospital, an expected average of 24 weeks.
  Each week the participant wears the accelerometers on both wrists during the 1 hour videotaping session, including 30-minute driving and 30-minute natural play. The accelerometers code the physical activity for driving and playing. Combining with the results from videotapes, this data enables us to understand the frequency and duration of bimanual use in different activities (i.e., manual exploration).

SECONDARY OUTCOMES:
Change from baseline in Body Function/Structure at 12 weeks and 24 weeks as assessed by 5-repetition Sit-to-stand (STS) test | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  A test that measures the time require to complete five consecutive sit-to-stand to-sit cycle as quickly as possible timed using a stop watch. Participants will be tested barefoot on a firm mat and the starting position with hip flexed at 90 degree and knee flexed at 105 degree. The ICCs of intra-session reliability and test-retest reliability were 0.95 and 0.99 respectively. The convergent validity was supported by significant correlation with isometric muscle strength, scores of Gross Motor Function Measure, and gait function (r or rho = 0.45-0.78).
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Bayley Scales of Development | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  The Bayley Scales of Development is an internationally recognized set of developmental tests that involve play and parental questionnaires. The Bayley has subsets of tests for motor (fine and gross), language (receptive and expressive), and cognitive development, ages from 0-3 years old.
Change from baseline in General Development at 12 weeks and 24 weeks as assessed by The Affordances in the Home Environment for Motor Development (AHEMD) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  AHEMD is a reliable and valid assessment to assess the quality and quantity of motor development opportunities in the home during early childhood. Age-related AHEMD questionnaires were developed (3-to-18 months; and 18-to-42 months) and translated into four different languages: English, Chinese Portuguese, and Spanish. Test-retest reliabilities for AHEMD-Toddler-C were adequate (0.46~0.93). For convergent validity, the correlation coefficients between AHEMD and HOME were 0.44.
Change from baseline in Participation level at 12 weeks and 24 weeks as assessed by The Goal Attainment Scale (GAS) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  GAS is a family-centered, criterion-referenced and responsive tool. There are 5 possible outcomes: a score of 0 means the child has attained the goal, whereas scores of -2 and -1 represent lower than expected performance and +1 and +2 are higher than expected performance. It has excellent inter-rater agreements with inter-class correlations of 0.90 or above. GAS was shown to correlate strongly with other measures that showed change, and it discriminated between lower and higher functional or QOL status.
Change from baseline in Parents' Perception at 12 weeks and 24 weeks as assessed by Parenting Stress Index (PSI) | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  PSI is a tool that was designed to measure the overall level of parenting stress experienced by parents of children between the ages of one month and twelve years. PSI showed very good reliability (from parent : .55-.80). The validity was well established (factorial validity: 41% of variance on child section accounted for by 6 factors; 44% on Parent section by 7 parent factors).
The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version | It will be administered a total of 3 times during the whole study, including the beginning and end of the 12-week intervention, and the end of the 12-week follow up.
  The Revised Dimensions of Mastery Questionnaire (DMQ 18) - Chinese version: was used to measure both instrumental and expressive aspects of mastery motivation by caregiver report. There are 7 scales (cognitive/object persistence, gross motor persistence, social mastery motivation with adults, social mastery motivation with children/peers, mastery pleasure, negative reactions to challenge in mastery situations, and general competence) and Likert-type items rated 1-5(from not at all like this child to exactly like this child). The DMQ 18 contained four parallel age-related versions for children aged 6 months to 19 years (infant, preschool, school-age rated by adults, and school-age self-report). The DMQ 18 show good internal consistency (.72-.96). The intra- and inter-rater reliability were acceptable for the DMQ18 (ICCs=0.61-0.87).

CONTACTS AND LOCATIONS:
Overall Officials: HsiangHan Huang, ScD, Principal Investigator — Chang Gung University
Locations (1):
- Chang Gung University, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Huang HH, Lee YT, Lai CL, Lin MC. On-time power mobility and physical activity in toddlers with motor delays: A randomized controlled trial using body-worn sensors. Assist Technol. 2025 Mar 4;37(2):111-119. doi: 10.1080/10400435.2024.2423606. Epub 2024 Nov 7. PMID 39508783
- [Derived] Huang HH, Tsai WY, Lin YN, Hung CY, Chan AT. Caregivers' Perceptions of Ride-On Cars and Behavioral Changes for Young Children With Motor Delays. Pediatr Phys Ther. 2024 Jan 1;36(1):42-51. doi: 10.1097/PEP.0000000000001066. Epub 2023 Oct 11. PMID 37820358